CLINICAL TRIAL: NCT04484987
Title: The Effect of Time-Restricted Eating in Cardiometabolic Health
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding withdrawn as the principal investigator moved from the USA to the UK
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1521859
Record Dates: First submitted 2020-07-17; First posted 2020-07-24 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2023-11

CONDITIONS: Obesity; Pre-diabetes
Keywords: Chrono-nutrition; Adipose tissue; Skeletal muscle; Insulin sensitivity; Diurnal rhythm
MeSH Terms: conditions — Obesity; Glucose Intolerance; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two diet interventions: TRE group (eating all their food for the day in 9 hours) or the control group (eating all their food for the day in 15 hours) for 12 weeks. Tests to asses changes in metabolism will be performed before and after the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TRE group (Other): Time-restricted eating group
  Interventions: Other: 9 hours daily eating window
- Control group (Other): Time-unrestricted eating group
  Interventions: Other: 15 hours daily eating window

INTERVENTIONS:
Other: 9 hours daily eating window — Participants assigned to the TRE group will have to consume all their daily meals and snacks during a 9-hour window for 12 weeks.
  Arms: TRE group
Other: 15 hours daily eating window — Participants assigned to the control group will have to consume all their daily meals and snacks during a 15-hour window for 12 weeks.
  Arms: Control group

SUMMARY:
Time-restricted eating (TRE) is a dietary manipulation that involves restricting food intake to 6-12 h/day with no energy intake the rest of the day. In rodents, TRE improves metabolic function without caloric restriction, potentially by activating nutrient sensing mechanisms and effects on circadian oscillations. However, an understanding of the effect of TRE on cardiometabolic health in people is not clear and few studies have evaluated this issue. Accordingly, the investigators propose to conduct a randomized controlled trial in people with obesity and prediabetes to determine the effect of 9 h TRE for 12 weeks, without a change in body weight, on key metabolic outcomes that are risk factors for cardiovascular disease (CVD): 1) multi-organ insulin sensitivity; 2) 24 h metabolic homeostasis and diurnal rhythm; and 3) adipose tissue and skeletal muscle biology. The proposed studies will elucidate the cardiometabolic implications of TRE in people with obesity and prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* body mass index 30-39.9 kg/m2
* fasting plasma glucose 100-125 mg/dl, or 2h OGTT plasma glucose 140-199 mg/dl or hemoglobin A1C 5.7-6.4%
* self-reported habitual eating period > 15 h per day

Exclusion Criteria:

* shift worker, recent or expected travel crossing time zones
* fasting >12 h/day more than once a week or vegan
* shift worker, recent or expected travel crossing time zones
* fasting >12 h/day more than once a week or vegan
* > once a week no food intake after 1800 h
* habitually waking up before 0400 h and sleeping before 2230 h
* ≥ 150 min per week of structured exercise
* unstable weight (>5% change the last 2 months)
* type 2 diabetes or other major chronic disease
* sleep disorder
* cancer in last 5 years
* conditions that render subject unable to complete all testing procedures
* use of medications that affect the study outcome measures or increase the risk of study procedures and that cannot be temporarily discontinued (e.g., steroids, alpha or beta adrenergic blockers or agonists, etc.)
* smoking and illegal drug use
* pregnant or lactating
* menopause
* individuals that have performed procedures involving substantial exposure to radiation in the last 12 months
* gastrointestinal or bariatric surgery
* unable to grant voluntary informed consent or comply with the study instructions
* individuals who are not yet adults (infants, children, teenagers)
* prisoners

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 3 months (pre-post intervention)
  Insulin sensitivity will be assessed by using a hyperinsulinemic euglycemic clamp procedure in conjunction with infusion of stable isotope tracers.
24 h glycemic control | 3 months (pre-post intervention)
  Changes in plasma glucose concentration will be assessed during a 24 h feeding study.
Adipose tissue gene expression | 3 months (pre-post intervention)
  Changes in the expression of genes involved in energy metabolism will be assessed by using qPCR.

SECONDARY OUTCOMES:
Peripheral diurnal rhythmicity in in peripheral mononuclear blood cells | 3 months (pre-post intervention)
  We will evaluate changes in clock gene expression

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will primarily include data collected specifically for the study, but it will also contain some demographic information and historical data regarding family history of diabetes, obesity, and cardiovascular disease. Upon publication of the primary manuscript, we will consider requests to make the study-related data and relevant demographic information (such as ethnicity) available to other investigators. The final dataset, which will not include subject names, will be further stripped of any other unique identifiers and prepared in accordance with all HIPAA regulations prior to release for sharing. No unique subject characteristics will be included in any reports generated by use of the data.
Supporting Information: Study Protocol
Time Frame: Upon publication of the study data.

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/a-study-of-time-restricted-eating-on-heart-health-metabolism-306499/